CLINICAL TRIAL: NCT05098028
Title: A Phase 2a Randomized, Double-Blind, Placebo-Controlled Study to Characterize the Pharmacokinetics and Pharmacodynamics of Rifaximin Novel Formulations in Patients With Sickle Cell Disease
Brief Title: Pharmacokinetics and Pharmacodynamics of Rifaximin Novel Formulations in Patients With Sickle Cell Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RBSC2161
Record Dates: First submitted 2021-10-18; First posted 2021-10-28 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Low Dose Rifaximin ER (Experimental): twice daily
  Interventions: Drug: Low Dose Rifaximin ER
- Low Dose Rifaximin DER (Experimental): twice daily
  Interventions: Drug: Low Dose Rifaximin DER
- High Dose Rifaximin ER (Experimental): twice daily
  Interventions: Drug: High Dose Rifaximin ER
- High Dose Rifaximin DER (Experimental): twice daily
  Interventions: Drug: High Dose Rifaximin DER
- Placebo (Placebo Comparator): twice daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Low Dose Rifaximin ER — Low Dose Rifaximin Extended Release Twice Daily
  Arms: Low Dose Rifaximin ER
Drug: Low Dose Rifaximin DER — Low Dose Rifaximin Delayed Extended Release Twice Daily
  Arms: Low Dose Rifaximin DER
Drug: High Dose Rifaximin ER — High Dose Rifaximin Extended Release Twice Daily
  Arms: High Dose Rifaximin ER
Drug: High Dose Rifaximin DER — High Dose Rifaximin Delayed Extended Release Twice Daily
  Arms: High Dose Rifaximin DER
Drug: Placebo — Placebo Twice Daily
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled study in sickle cell disease participants with a history of Vaso-occlusive Crises (VOCs). Approximately 60 participants with sickle cell disease will be enrolled and randomized: 12 participants in each of four active novel formulation rifaximin groups and 6 participants in each of 2 placebo groups.

ELIGIBILITY:
Inclusion Criteria:

1. ability and willingness to sign a written informed consent form.
2. between the ages of 18 to 70 years old (inclusive) at the time of consent.
3. SCD of any genotype (HbSS, HbSC, HbS β-thalassemia). If the subject's genotype has not been previously documented, genotyping will be performed during Screening using high-performance liquid chromatography (HPLC)/electrophoresis.
4. least 2 VOCs within the 12 months prior to Screening.
5. if receiving hydroxyurea (HU)/hydroxycarbamide (HC), subject must have been receiving the treatment for at least 6 months prior to Screening and must agree to maintain the same dose and schedule for the duration of the study.
6. must have laboratory values at Screening as follows:

   1. Absolute Neutrophil Count ≥1.0 x 109/L
   2. Platelets ≥ 75 x 109/L
   3. Hemoglobin (Hgb) ≥ 6.0 g/dL
   4. Glomerular filtration rate (GFR) ≥ 45 mL/min/1.73 m2 using the CKD-EPI formula
   5. Total bilirubin ≤ 15 mg/dL
   6. Alanine transaminase (ALT) ≤ 3.0 x ULN
   7. International Normalized Ratio (INR) ≤ 2.0
7. Eastern Cooperate Oncology Group (ECOG) performance status ≤ 2
8. Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, must have a negative serum pregnancy test at Screening and agree to use standard prevention methods for the duration of the study.

Exclusion Criteria:

1. receiving concomitant treatment with voxelotor, crizanlizumab, or L-glutamine.
2. any history of stem cell transplant, is planning to begin or has received in past 30 days.
3. acute VOC, requiring a visit to a medical facility and/or healthcare professional, ending within 7 days prior to Day 1 dosing.
4. has received any blood products within 30 days prior to Day 1 dosing.
5. uncontrolled liver disease or renal impairment, ulcerative colitis, Crohn's disease, or other chronic GI disorder.
6. has received active treatment in another investigational trial within 30 days or 5 half-lives of the last dose of the investigational agent, whichever is greater, prior to Screening.
7. has received penicillin prophylaxis or antibiotics for treatment of infection within 30 days or 5 half-lives of the treatment, whichever is greater, prior to Screening.
8. significant medical condition that required hospitalization (other than for a VOC) within 2 months prior to Screening.
9. planning on undergoing an exchange transfusion during the duration of the study or has completed one within 4 weeks prior to Day 1 dosing.
10. hypersensitivity to rifaximin, rifampin, rifamycin antimicrobial agents, or any components of rifaximin ER and DER.
11. pregnant or a nursing woman.
12. history of illicit drug use or abuse, either documented or in the opinion of the Investigator.
13. using any medication that is known to inhibit or induce CYP3A4, or P-gp and OATP1B1/B3 within 30 days or 5 half-lives, whichever is longer, prior to Day 1 dosing, or in the opinion of the Investigator, may affect the evaluation of the study product or place the subject at undue risk.
14. has had any prior gastrointestinal surgery which has altered the anatomy of the esophagus, stomach, or small/large intestine (with the exception of appendectomy, cholecystectomy, and fundoplication).
15. has had a colonoscopy or sigmoidoscopy within 30 days prior to Day 1 or plans to undergo such a procedure during the duration of the study.
16. has used bowel prep, laxative, or enema within 30 days prior to Day 1.
17. bleeding disorder including, but not limited to, acquired or congenital platelet function defects, disseminated intravascular coagulation (DIC), bleeding factor deficiencies, hemophilia, idiopathic thrombocytopenia purpura (ITP), or von Willebrand's disease.
18. planning to undergo a major surgical procedure during the duration of the study.
19. positive test for human immunodeficiency virus (HIV)1 or HIV2.
20. active Hepatitis B infection (HBsAg positive). Prior infection that is not active (i.e., HBsAg negative, HBcAb positive, and HBsAb positive) is permitted.
21. positive test for Hepatitis C (HCV RNA). Prior infection with spontaneous resolution or sustained resolution for ≥ 24 weeks after cessation of antivirals is permitted.
22. active COVID-19 infection or complication(s) related to COVID 19 infection that are unresolved or, in the opinion of the Investigator, may affect evaluation of the study drug or place the subject at undue risk.
23. received a vaccine (including COVID-19 vaccine) within 2 weeks prior to Screening. If subject has received their first of two COVID-19 vaccination doses, as applicable, they must wait for at least 2 weeks after receiving the second dose, and be symptom-free, prior to beginning Screening. Subject must not be planning for COVID-19 or other vaccinations while on study.
24. malignant disease. Exceptions include malignancies that were treated curatively and have not recurred within 2 years prior to study treatment, completely resected basal cell and squamous cell skin cancers, and any completely resected carcinoma in situ.
25. prolonged QT interval as assessed by ECG history within the past 3 months. For subjects with no historical ECG information, subject has a resting QTcF ≥ 460 msec for males and ≥ 470 msec for females at Screening.
26. any unstable cardiac condition that, in the opinion of the Investigator, may worsen during the study or interfere with successful evaluation of the study treatment.
27. serious mental or physical illness which, in the opinion of the Investigator, would compromise participation in the study.
28. any condition which, in the opinion of the Investigator, is likely to interfere with the successful collection of the measurements required for the study.
29. unable to understand or comply with study instructions and requirements.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2022-03-22 (Actual); Primary Completion 2023-09-04 (Actual); Study Completion 2023-09-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Varsha Bhatt, Study Director — Bausch Health
Locations (8):
- United States (5):
  - Bausch Site 105, Orange, California
  - Bausch Site 103, Denver, Colorado
  - Bausch Site 104, Atlanta, Georgia
  - Bausch Site 101, Syracuse, New York
  - Bausch Site 102, Greenville, North Carolina
- Bausch Site 201, Montreal, Quebec, Canada
- Kenya (2):
  - Bausch Site 501, Eldoret
  - Bausch Site 502, Kisumu

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Low Dose Rifaximin ER | High Dose Rifaximin ER | Low Dose Rifaximin DER | High Dose Rifaximin DER | Placebo
Started | 7 | 8 | 11 | 9 | 9
Completed | 7 | 8 | 11 | 9 | 8
Not Completed | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Low Dose Rifaximin ER | High Dose Rifaximin ER | Low Dose Rifaximin DER | High Dose Rifaximin DER | Placebo | Total
Number analyzed (Participants) | 7 | 8 | 11 | 9 | 9 | 44
Age, Continuous [Mean (Standard Deviation); unit: years] | 23.0 (3.74) | 24.6 (4.17) | 29.3 (10.54) | 22.6 (4.16) | 25.8 (5.93) | 25.3 (6.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 8 | 2 | 3 | 23
  Male | 2 | 3 | 3 | 7 | 6 | 21
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 6 | 7 | 10 | 7 | 7 | 37
  White | 1 | 0 | 1 | 1 | 1 | 4
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 1 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Maximum Plasma Concentration
Description: Maximum observed plasma concentration
Time Frame: Day 29
Population: Pharmacokinetic population included all participants who took at least 1 dose of active study treatment and had at least 1 blood sample collected and analyzed for at least 1 quantifiable plasma concentration for rifaximin and/or 25-desacetyl rifaximin without significant protocol violations or events with potential to affect the PK concentrations.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Low Dose Rifaximin ER | High Dose Rifaximin ER | Low Dose Rifaximin DER | High Dose Rifaximin DER | Placebo
Number analyzed (Participants) | 5 | 6 | 7 | 5 | 0
ng/mL | 0.5835 (86.3) | 0.7425 (58.4) | 0.2186 (124.0) | 0.7128 (50.1) |

ADVERSE EVENTS:
Time Frame: 28 days of treatment and 2 weeks of follow-up.
Arm/Group | Low Dose Rifaximin ER | High Dose Rifaximin ER | Low Dose Rifaximin DER | High Dose Rifaximin DER | Placebo
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/8 | 0/11 | 0/9 | 0/9
Serious Adverse Events (participants affected / at risk) | 1/7 | 0/8 | 2/11 | 1/9 | 0/9
Other Adverse Events (participants affected / at risk) | 7/7 | 8/8 | 9/11 | 8/9 | 5/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Low Dose Rifaximin ER (N=7) | High Dose Rifaximin ER (N=8) | Low Dose Rifaximin DER (N=11) | High Dose Rifaximin DER (N=9) | Placebo (N=9)
Anemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 1 | 0
Malaria (Infections and infestations) | 1 | 0 | 1 | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 1 | 1 | 0
Sepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Abortion complete (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Low Dose Rifaximin ER (N=7) | High Dose Rifaximin ER (N=8) | Low Dose Rifaximin DER (N=11) | High Dose Rifaximin DER (N=9) | Placebo (N=9)
Anemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
Hypochromic anemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0
Iron deficiency anemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0
Thrombocytosis (Blood and lymphatic system disorders) | 2 | 2 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1
Eye pruritus (Eye disorders) | 0 | 0 | 1 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 4 | 3 | 4 | 0 | 3
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 1
Diarrhea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Hyperchlorhydria (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 1 | 1 | 1 | 2
Vessel puncture site pain (General disorders) | 0 | 0 | 0 | 0 | 2
Non-cardiac chest pain (General disorders) | 1 | 1 | 1 | 2 | 1
Chills (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Puncture site pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Swelling face (General disorders) | 0 | 0 | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 1 | 0 | 0
Portal fibrosis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0
Bacterial infection (Infections and infestations) | 2 | 2 | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Malaria (Infections and infestations) | 1 | 0 | 0 | 1 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Body tinea (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Fungal skin infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Lip infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Septic rash (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Tinea versicolour (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 1 | 0 | 0
Vulvovaginal candidiasis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
White blood cell count increased (Investigations) | 1 | 1 | 0 | 0 | 2
Neutrophil count increased (Investigations) | 1 | 0 | 0 | 0 | 1
Urine leukocyte esterase positive (Investigations) | 1 | 1 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 1 | 1 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 1 | 1 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 0 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 1 | 0 | 0 | 0
Blood lactate dehydrogenase increased (Investigations) | 1 | 1 | 1 | 0 | 0
Urine blood present (Investigations) | 0 | 0 | 0 | 1 | 0
C-reactive protein increased (Investigations) | 0 | 2 | 1 | 0 | 0
High density lipoprotein decreased (Investigations) | 1 | 0 | 0 | 0 | 0
Lymphocyte count increased (Investigations) | 1 | 0 | 0 | 0 | 0
Nitrite urine present (Investigations) | 1 | 0 | 1 | 1 | 0
Platelet count decreased (Investigations) | 0 | 0 | 1 | 0 | 0
Platelet count increased (Investigations) | 2 | 0 | 0 | 0 | 0
Streptococcus test positive (Investigations) | 0 | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 1 | 1 | 3 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 4 | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 4 | 4 | 3 | 3 | 2
Dizziness (Nervous system disorders) | 0 | 1 | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Urine abnormality (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Dysmenorrhea (Reproductive system and breast disorders) | 0 | 1 | 1 | 0 | 0
Ovarian cyst (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0
Vulvovaginal rash (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Please contact sponsor for details.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-04-12): https://cdn.clinicaltrials.gov/large-docs/28/NCT05098028/Prot_SAP_000.pdf